CLINICAL TRIAL: NCT07343206
Title: Efficacy of Early Norepinephrine Administration and Rapid Dose Adjustment in Adult Septic Shock Patients: A Multicenter Randomized Controlled Trial
Brief Title: Early Norepinephrine Administration and Rapid Dose Adjustment
Acronym: CENSER2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Maharaj Nakorn Si Thammarat (Unknown); Kalasin Hospital (Other); Khon Kaen Hospital (Other Government); Udon Thani Regional Hospital (Unknown); Hat Yai Hospital (Unknown)
Responsible Party: Principal Investigator, Wasin Pansiritanachot, Lecturer, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 930/2025
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Septic Shock
Keywords: septic shock; norepinephrine; sepsis; hypotension
MeSH Terms: conditions — Sepsis; Shock, Septic; Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Norepinephrine 4 mg in 250 mL D5W, initiated at 0.05 mcg/kg/min. Titrate by 0.025 mcg/kg/min every 15 minutes if MAP <65 mmHg, up to 0.15 mcg/kg/min maximum. Rescue norepinephrine available if needed (separate line). Limb ischemia monitoring every 15 minutes.
  Duration: 24 hours.
  Interventions: Drug: Early norepinephrine administration and rapid dose adjustment
- Control (Sham Comparator): Placebo (D5W 250 mL) with an identical dosing schedule. Rescue norepinephrine available via a separate line. Same monitoring protocols.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Early norepinephrine administration and rapid dose adjustment — Norepinephrine 4 mg in 250 mL D5W, initiated at 0.05 mcg/kg/min. Titrate by 0.025 mcg/kg/min every 15 minutes if MAP <65 mmHg, up to 0.15 mcg/kg/min maximum. Rescue norepinephrine available if needed (separate line). Limb ischemia monitoring every 15 minutes.
  Duration: 24 hours.
  Arms: Intervention
Drug: Control — Placebo (D5W 250 mL) with an identical dosing schedule. Rescue norepinephrine available via a separate line. Same monitoring protocols.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to determine whether early initiation of norepinephrine with rapid dose adjustment improves clinical outcomes in adult patients with septic shock. The study aims to evaluate the effect of early norepinephrine administration on mortality, hemodynamic stabilization, and resuscitation efficiency in adults aged 18 years and older diagnosed with septic shock.

The main questions it aims to answer are:

* Does early norepinephrine administration with rapid dose titration reduce 28-day mortality compared with standard treatment?
* Does early norepinephrine administration with rapid dose tiration lead to faster shock control and reduced fluid requirements without increasing treatment-related adverse events?

Researchers will compare early norepinephrine administration with rapid dose adjustment to placebo with standard sequential resuscitation and rescue norepinephrine as needed to see if early vasopressor initiation improves survival, shock resolution, and safety outcomes.

Participants will:

* Receive either norepinephrine or placebo infusion initiated within one hour of septic shock diagnosis, with dose adjustment every 15 minutes according to a standardized protocol
* Undergo close hemodynamic and safety monitoring, including frequent vital sign assessment and limb perfusion evaluation
* Receive standard sepsis care, including fluid resuscitation, antibiotics, and organ support as clinically indicated
* Be followed for clinical outcomes and adverse events for up to 28 days after enrollment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sepsis: SOFA ≥2 with suspected infection
* Mean arterial pressure <65 mmHg
* Diagnosed within 3 hours

Exclusion Criteria:

* Do-not-resuscitate orders
* Pregnancy
* Severe concurrent conditions (acute stroke, acute coronary syndrome, acute pulmonary edema, status asthmaticus, active gastrointestinal bleeding, status epilepticus, severe burn, severe trauma, and fatal drug overdose, End-stage malignancy
* Peripheral arterial disease
* Prior norepinephrine administration
* Recurrent shock in the same patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
28-day survival | From enrollment to 28 days after enrollment
  Survival at 28-day after enrollment. Telephone follow-up for patients who are discharged before 28 days.

SECONDARY OUTCOMES:
Number of participants with shock control achieved | From enrollment to 6 hours after enrollment
  Shock control defined as mean arterial pressure greater than 65 mmHg combined with urine output greater than 0.5 milliliters per kilogram per hour OR lactate clearance greater than 10 percent within 6 hours
Duration of intensive care unit stay | From enrollment to hospital discharge or 90 days (whichever comes first)
  Days of intensive care unit stay
Duration of hospital stay | From enrollment to hospital discharge or 90 days (whichever comes first)
  Days of hospital stay
Duration of mechanical ventilation | From enrollment to hospital discharge or 90 days (whichever comes first)
  Days on mechanical ventilation, including endotracheal tube and tracheostomy
Duration of renal replacement therapy | From enrollment to hospital discharge or 90 days (whichever comes first)
  Days requiring renal replacement therapy, including continuous renal replacement therapy, intermittent hemodialysis, and peritoneal dialysis, that is newly initiated during this admission. Maintaining chronic hemodialysis is excluded.
Duration of vasopressor therapy | From enrollment to hospital discharge or 90 days (whichever comes first)
  Days requiring vasopressor therapy
Time to Achievement of Early Goal-Directed Therapy Targets | From study drug initiation until achievement of all EGDT targets or up to 6 hours
  Time in hours to achieve ALL EGDT targets: MAP ≥65 mmHg, urine output ≥0.5 mL/kg/hr, lactate clearance ≥10%, and ScvO₂ ≥70% (when measured)
Cumulative Fluid Volume Administered | Multiple assessments at: - Before randomization (baseline) - 1 hour after study drug initiation - 6 hours after study drug initiation - 24 hours (Day 1) 48 hours (Day 2) 72 hours (Day 3) after study drug initiation
  Total volume in milliliters of intravenous crystalloid and colloid fluids administered during first 24 hours and first 72 hours Time Frame: At 1 hour, 6 hours, 24 hours (Day 1), 48 hours (Day 2), and 72 hours (Day 3) after treatment initiation
Incidence of Pulmonary Edema | From diagnosis until hospital discharge 90 days or death
  New-onset cardiogenic pulmonary edema or non-cardiogenic pulmonary edema
Treatment-Related Adverse Events Including Cardiac Arrhythmias | From study drug initiation until hospital discharge or death, assessed 90 days
  Composite outcome including new-onset arrhythmias (AF, AFL, SVT, VT, VF, AV block, bradycardia), limb/mesenteric ischemia, skin necrosis, and severe hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Permpikul, Professor, Principal Investigator — Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (6):
- Thailand (6):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Kalasin Hospital, Kalasin, Changwat Kalasin
  - Khon Kaen hospital, Khon Kaen, Changwat Khon Kaen
  - Udon Thani Hospital, Udon Thani, Changwat Udon Thani
  - Hatyai Hospital, Hat Yai, Hat Yai
  - Maharaj Nakhon Si Thammarat Hospital, Nakhon Si Thammarat, ์Nakhon Si Thammarat

IPD SHARING:
Plan to Share IPD: Undecided
De-identified anonymized patient data will be available upon reasonable request.